CLINICAL TRIAL: NCT01777334
Title: A Multicenter, Trial Comparing the Efficacy and Safety of Umeclidinium/Vilanterol 62.5/25 mcg Once Daily With Tiotropium 18 mcg Once Daily Over 24 Weeks in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: The Purpose of This Study is to Evaluate the Spirometric Effect (Trough FEV1) of Umeclidinium/Vilanterol 62.5/25 mcg Once Daily Compared With Tiotriopium 18 mcg Once Daily Over a 24-week Treatment Period in Subjects With COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 117115
Record Dates: First submitted 2013-01-24; First posted 2013-01-28 (Estimated); Results first posted 2014-06-05 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — GSK573719; vilanterol; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Umeclidinium/Vilanterol (Experimental): Long-acting muscarinic antagonist (LAMA)/Long-acting Beta agonist (LABA)
  Interventions: Drug: Umeclidinium/Vilanterol 62.5/25 mcg
- Tiotropium (Active Comparator): Long-acting muscarinic antagonist (LAMA)
  Interventions: Drug: Tiotropium 18 mcg

INTERVENTIONS:
Drug: Umeclidinium/Vilanterol 62.5/25 mcg — Inhalation Powder
  Arms: Umeclidinium/Vilanterol
Drug: Tiotropium 18 mcg — Inhalation Powder
  Arms: Tiotropium

SUMMARY:
The purpose of this 24 week study is to evaluate the spirometric lung function effect (trough FEV1) of Umeclidinium/Vilanterol 62.5/25 once daily compared to Tiotropium 18 mcg once daily along with safety assessments in subjects with COPD.

DETAILED DESCRIPTION:
This is a Phase IIIb multicenter, randomized, double-dummy, parallel group study to evaluate the efficacy and safety of UMEC/VI Inhalation Powder (62.5/25 mcg) when administered once-daily via a novel dry powder inhaler (DPI) compared with tiotropium (18 mcg) administered once-daily via the HandiHaler over a treatment period of 24 weeks in subjects with COPD. Eligible subjects will be randomized 1:1 to UMEC/VI Inhalation Powder (62.5/25 mcg), or tiotropium (18 mcg) for 24 weeks.

There will be a total of 10 study clinic visits conducted on an outpatient basis. Subjects who meet the eligibility criteria at Screening (Visit 1) will complete a 7- to 10-day run-in period followed by a 24-week treatment period. Clinic visits will be at Screening, Randomization (Day 1), Day 2 and after 4, 8, 12, 16, 20 and 24 weeks, and 1 day after the Week 24 visit (Visit 1 to Visit 10, respectively). Additionally a safety Follow-Up assessment will be conducted either by phone call or clinic visit where required approximately 7 days after the end of the study treatment (Visit 10 or Early Withdrawal, if applicable). The total duration of subject participation, including the Follow-Up will be approximately 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Type of subject: Outpatient.
* Informed Consent: A signed and dated written informed consent prior to study participation.
* Age: Subjects 40 years of age or older at Visit 1.
* Gender: Male or female subjects.

A female is eligible to enter and participate in the study if she is of:

Non-child bearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is post-menopausal or surgically sterile). Surgically sterile females are defined as those with a documented hysterectomy and/or bilateral oophorectomy or tubal ligation. Post-menopausal females are defined as being amenorrhoeic for greater than 1 year with an appropriate clinical profile, e.g. age appropriate, > 45 years, in the absence of hormone replacement therapy.

OR

Child bearing potential, has a negative pregnancy test at screening, and agrees to one of the following acceptable contraceptive methods used consistently and correctly (i.e. in accordance with the approved product label and the instructions of the physician for the duration of the study - screening to follow-up contact):

* Abstinence
* Oral Contraceptive, either combined or progestogen alone
* Injectable progestogen
* Implants of levonorgestrel
* Estrogenic vaginal ring
* Percutaneous contraceptive patches
* Intrauterine device (IUD) or intrauterine system (IUS) that meets the SOP effectiveness criteria as stated in the product label
* Male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study, and this male is the sole partner for that subject. For this definition, "documented" refers to the outcome of the investigator's/designee's medical examination of the subject or review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records.
* Double barrier method: condom and an occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/film/cream/suppository)

  * COPD Diagnosis: An established clinical history of COPD in accordance with the definition by the American Thoracic Society/European Respiratory Society [Celli, 2004].
  * Smoking History: Current or former cigarette smokers with a history of cigarette smoking of >=10 pack-years [number of pack years = (number of cigarettes per day / 20) x number of years smoked (e.g., 20 cigarettes per day for 10 years, or 10 cigarettes per day for 20 years)]. Previous smokers are defined as those who have stopped smoking for at least 6 months prior to Visit 1.

Note: Pipe and/or cigar use cannot be used to calculate pack-year history

* Severity of Disease: A pre and post-albuterol/salbutamol FEV1/FVC ratio of <0.70 and a pre and post-albuterol/salbutamol FEV1 of FEV1 of <=70% of predicted normal values calculated using NHANES III reference equations at Visit 1 [Hankinson, 1999; Hankinson, 2010].
* Dyspnea: A score of ≥2 on the Modified Medical Research Council Dyspnea Scale (mMRC) at Visit 1.

Exclusion Criteria:

* Pregnancy: Women who are pregnant or lactating or are planning on becoming pregnant during the study.
* Asthma: A current diagnosis of asthma.
* Other Respiratory Disorders: Known alpha 1 antitrypsin deficiency, active lung infections (such as tuberculosis), and lung cancer are absolute exclusionary conditions. A subject who, in the opinion of the investigator, has any other significant respiratory conditions in addition to COPD should be excluded. Examples may include clinically significant bronchiectasis, pulmonary hypertension, sarcoidosis, or interstitial lung disease.
* Other Diseases/Abnormalities: Subjects with historical or current evidence of clinically significant cardiovascular, neurological, psychiatric, renal, hepatic, immunological, endocrine (including uncontrolled diabetes or thyroid disease) or hematological abnormalities that are uncontrolled and/or a previous history of cancer in remission for <5 years prior to Visit 1 (localized carcinoma of the skin that has been resected for cure is not exclusionary). Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the subject at risk through participation, or which would affect the efficacy or safety analysis if the disease/condition exacerbated during the study.
* Contraindications: A history of allergy or hypersensitivity to any anticholinergic/muscarinic receptor antagonist, beta2-agonist, lactose/milk protein or magnesium stearate or a medical condition such as narrow-angle glaucoma, prostatic hypertrophy or bladder neck obstruction that, in the opinion of the study physician contraindicates study participation or use of an inhaled anticholinergic.
* Hospitalization: Hospitalization for COPD or pneumonia within 12 weeks prior to Visit 1.
* Lung Resection: Subjects with lung volume reduction surgery within the 12 months prior to Screening (Visit 1).
* 12-Lead ECG: An abnormal and significant ECG finding from the 12-lead ECG conducted at Visit 1, including the presence of a paced rhythm on a 12-lead electrocardiogram (ECG) which causes the underlying rhythm and ECG to be obscured. Investigators will be provided with ECG reviews conducted by a centralized independent cardiologist to assist in evaluation of subject eligibility. Specific ECG findings that preclude subject eligibility are listed in Appendix 4. The study investigator will determine the medical significance of any ECG abnormalities not listed in Appendix 4.
* Medication Prior to Spirometry: Unable to withhold albuterol/salbutamol for the 4 hour period required prior to spirometry testing at each study visit.
* Use of certain medications according to defined time intervals prior to Screening (Visit 1).
* Oxygen: Use of long-term oxygen therapy (LTOT) described as oxygen therapy prescribed for greater than 12 hours a day. As-needed oxygen use (i.e., >=12 hours per day) is not exclusionary.
* Nebulized Therapy: Regular use (prescribed for use every day, not for as-needed use) of short-acting bronchodilators (e.g., albuterol/salbutamol) via nebulized therapy.
* Pulmonary Rehabilitation Program: Participation in the acute phase of a pulmonary rehabilitation program within 4 weeks prior to Visit 1. Subjects who are in the maintenance phase of a pulmonary rehabilitation program are not excluded.
* Drug or Alcohol Abuse: A known or suspected history of alcohol or drug abuse within 2 years prior to Visit 1.
* Affiliation with Investigator Site: Is an investigator, sub-investigator, study coordinator, employee of a participating investigator or study site, or immediate family member of the aforementioned that is involved in this study.
* Previous use of study drug: Previous participation in DB2113360 or DB2113374.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 905 (Actual)
Dates: Start 2013-01-23 (Actual); Primary Completion 2013-09-24 (Actual); Study Completion 2013-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (61):
- United States (17):
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, Panama City, Florida
  - GSK Investigational Site, Coeur d'Alene, Idaho
  - GSK Investigational Site, Saint Charles, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Easley, South Carolina
  - GSK Investigational Site, Gaffney, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Rock Hill, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Union, South Carolina
  - GSK Investigational Site, Johnson City, Tennessee
- GSK Investigational Site, Ciudad Autnónoma de Buenos Aires, Buenos Aires, Argentina
- Bulgaria (7):
  - GSK Investigational Site, Dimitrovgrad
  - GSK Investigational Site, Pleven
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Rousse
  - GSK Investigational Site, Stara Zagora
  - GSK Investigational Site, Troyan Municipality
  - GSK Investigational Site, Varna
- Canada (9):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Moncton, New Brunswick
  - GSK Investigational Site, Burlington, Ontario
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Saint-Charles-Borromée, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
- Germany (7):
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Neu-Isenburg, Hesse
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Geesthacht, Schleswig-Holstein
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Hungary (6):
  - GSK Investigational Site, Balassagyarmat
  - GSK Investigational Site, Budaörs
  - GSK Investigational Site, Debrecen
  - GSK Investigational Site, Gödöllő
  - GSK Investigational Site, Nyíregyháza
  - GSK Investigational Site, Szikszó
- Romania (4):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Codlea
  - GSK Investigational Site, Deva
- Russia (6):
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Belgorod
  - GSK Investigational Site, Krasnodar
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Pyatigorsk
  - GSK Investigational Site, Saint Petersburg
- Spain (4):
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Mérida (Badajoz)
  - GSK Investigational Site, Salt (gerona)
  - GSK Investigational Site, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Maleki-Yazdi MR, Singh D, Anzueto A, Tombs L, Fahy WA, Naya I. Assessing Short-term Deterioration in Maintenance-naive Patients with COPD Receiving Umeclidinium/Vilanterol and Tiotropium: A Pooled Analysis of Three Randomized Trials. Adv Ther. 2017 Jan;33(12):2188-2199. doi: 10.1007/s12325-016-0430-6. Epub 2016 Oct 28. PMID 27796912
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 117115 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 117115 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 117115 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 117115 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 117115 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 117115 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 117115 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants (par.) who met the eligibility criteria at Screening (Visit 1) completed a 7- to 10-day Run-in Period and entered a 24-week Treatment Period. 1191 par. signed the informed consent form and were assigned subject numbers, 1053 par. were screened and 905 par. were randomized and received at least one dose of study medication.
Groups:
- UMEC/VI 62.5/25 µg: Participants received umeclidinium bromide/vilanterol (UMEC/VI) 62.5/25 micrograms (µg) once daily (QD) each morning via a dry powder inhaler (DPI) and placebo QD each morning via a DPI for 24 weeks.
- TIO 18 µg: Participants received tiotropium (TIO) 18 µg QD each morning via a DPI and placebo QD each morning via a DPI for 24 weeks.
Period: Overall Study
Arm/Group | UMEC/VI 62.5/25 µg | TIO 18 µg
Started | 454 | 451
Completed | 401 | 388
Not Completed | 53 | 63
Not completed — Adverse Event | 18 | 14
Not completed — Lack of Efficacy | 15 | 29
Not completed — Protocol Violation | 3 | 7
Not completed — Lost to Follow-up | 3 | 2
Not completed — Withdrawal by Subject | 14 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | UMEC/VI 62.5/25 µg | TIO 18 µg | Total
Number analyzed (Participants) | 454 | 451 | 905
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.9 (8.41) | 62.7 (8.50) | 62.3 (8.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 144 | 148 | 292
  Male | 310 | 303 | 613
Race/Ethnicity, Customized [Number; unit: Participants]
  White/Caucasian/European Heritage | 438 | 442 | 880
  African American/African Heritage | 13 | 7 | 20
  American Indian or Alaska Native | 1 | 1 | 2
  White - Arabic/North African Heritage | 1 | 0 | 1
  Mixed Race | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (BL) in Trough Forced Expiratory Volume in One Second (FEV1) on Day 169 (Week 24)
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Trough FEV1 measurements were taken electronically by spirometry on Days 2, 28, 56, 84, 112, 140, 168, and 169. Baseline is defined as the mean of the assessments made 30 minutes (min) pre-dose and 5 min pre-dose on Treatment Day 1. Trough FEV1 is defined as the mean of the FEV1 values obtained at 23 and 24 hours (hr) after the previous morning's dosing (ie., trough FEV1 on Day 169 is the mean of the FEV1 values obtained 23 and 24 hr after the morning dosing on Day 168). Change from Baseline at a particular visit was calculated as the trough FEV1 value at that visit minus the Baseline value. Analysis was performed using a repeated measures model with covariates of treatment, Baseline (mean of the two assessmentsmade 30 min and 5 min pre-dose on Day 1), smoking status, center group, day, and day by Baseline and day by treatment interactions.
Time Frame: Baseline and Day 169
Population: Intent-to-Treat (ITT) Population: all participants randomized to treatment who received at least one dose of randomized study drug during the Treatment Period. Par. analyzed are those with data available at the presented time point; but, all par. without missing covariate information and with >=1 post-BL measurement were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | UMEC/VI 62.5/25 µg | TIO 18 µg
Number analyzed (Participants) | 400 | 388
Liters | 0.205 (0.0114) | 0.093 (0.0115)
Statistical Analysis 1: Comparison: UMEC/VI 62.5/25 µg vs TIO 18 µg; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.112, 95% CI 2-sided [0.081 to 0.144] — Least squares mean difference=UMEC/VI 62.5/25 µg minus TIO 18 µg

2. Secondary Outcome: Change From Baseline (BL) in Weighted Mean (WM) 0-6 Hour FEV1 Obtained Post-dose at Day 168
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. The WM FEV1 was derived by calculating the area under the FEV1/time curve (AUC) using the trapezoidal rule, and then dividing the value by the time interval over which the AUC was calculated. The WM was calculated at Days 1, 84, and 168 using the 0-6-hour post-dose FEV1 measurements collected on that day, which included pre-dose (Day 1: 30 minutes [min] and 5 min prior to dosing; other serial visits: 23 and 24 hours after the previous morning dose) and post-dose at 15 min, 30 min, 1 hour, 3 hours, and 6 hours. Change from BL at a particular visit was calculated as the WM value at that visit minus the BL value. Analysis was performed using a repeated measures model with covariates of treatment, BL (mean of the two assessments made 30 min and 5 min pre-dose on Day 1), smoking status, center group, day, and day by BL and day by treatment interactions.
Time Frame: Baseline and Day 168
Population: ITT Population. Par. analyzed are those with data available at the presented time point; but, all par. without missing covariate information and with >=1 post-Baseline measurement were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | UMEC/VI 62.5/25 µg | TIO 18 µg
Number analyzed (Participants) | 404 | 387
Liters | 0.276 (0.0124) | 0.170 (0.0126)

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious AEs were collected from the start of study medication until the end of treatment (up to 24 weeks).
Description: SAEs and non-serious AEs are reported for members of the ITT Population, comprised of all participants randomized to treatment who received at least one dose of randomized study drug during the Treatment Period.
Arm/Group | UMEC/VI 62.5/25 µg | TIO 18 µg
Serious Adverse Events (participants affected / at risk) | 16/454 | 17/451
Other Adverse Events (participants affected / at risk) | 71/454 | 72/451
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UMEC/VI 62.5/25 µg (N=454) | TIO 18 µg (N=451)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2
Appendicitis (Infections and infestations) | 1 | 0
Epiglottitis (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 1 | 0
Sudden death (General disorders) | 0 | 1
Arterial restenosis (Injury, poisoning and procedural complications) | 0 | 1
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Mental disorder (Psychiatric disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | UMEC/VI 62.5/25 µg (N=454) | TIO 18 µg (N=451)
Headache (Nervous system disorders) | 40 | 31
Nasopharyngitis (Infections and infestations) | 28 | 30
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.